CLINICAL TRIAL: NCT04658225
Title: Gingivitis Treated With Chlorhexidine 0.12% Mouthwash in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Gabriela Alessandra da Cruz Galhardo Camargo, Clinical Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE: 69912817.0.0000.5626.
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Age Problem
Keywords: Gingivitis; Periodontal treatment
MeSH Terms: conditions — Gingivitis | interventions — Chlorhexidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Thirty patients with gingivitis ages18 to 30 year with a probing depth of at most 3 mm and at least 20 teeth will select and evaluate at baseline and after 4 weeks. The periodontal clinical parameters will verify: plaque index (PI), gingival index (GI) and Simplified Oral Hygiene Index (OHIS). After evaluation of the clinical parameters, the patients will randomly allocated into two groups of 15 individuals to rinse with antimicrobials twice a day for a period of four weeks. Group A, received 0.12% chlorhexidine antimicrobian in a vial previously identified as solution 1 and group B, received saline solution identified as solution 2.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant will receiver mouthwash solution with labeled number, they will not know which solution will inside.
  Care provider - The research that will collect clinical parameter wil be different for researcher that will do the treatment.
  Investigator will not have contact with treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solution 1 (Active Comparator): 0.12% chlorhexidine
  Interventions: Procedure: 0.12% chlorhexidine
- Solution 2 (Placebo Comparator): Saline solution
  Interventions: Procedure: 0.12% chlorhexidine

INTERVENTIONS:
Procedure: 0.12% chlorhexidine — the patients were randomly allocated into two groups of 15 individuals to rinse with antimicrobials twice a day for a period of four weeks. Group A, received 0.12% chlorhexidine antimicrobian in a vial previously identified as solution 1 and group B, received saline solution identified as solution 2.
  Other Names: Saline Solution

SUMMARY:
The aim of this study will evaluate the effectiveness of 0.12% chlorhexidine solution as an anti-inflammatory agent and reducing the presence of biofilm in young adults.

DETAILED DESCRIPTION:
Thirty patients with gingivitis ages 18 to 30 year with a probing depth of at most 3 mm and at least 20 teeth will be selected and evaluate at baseline and after 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Presence of gingivitis
* Probing depth (PD) with maximum 3 mm
* Minimum of 20 teeth
* Age between 18 and 30 years old

Exclusion Criteria:

* Patients with periodontal disease (PD ≥ 4mm with clinical attachment loss)
* Diabetes
* Osteoporosis
* Pregnant or lactating females
* Smokers
* Users of immune suppressive medication
* Phenytoin or cyclosporine
* Calcium channel blockers
* Antibiotics
* Nonsteroidal anti-inflammatory drugs
* HIV+ or AIDS

Ages: 30 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Plaque Index | 30 days
  Check the biofilm as Ainano & Bay 1975 index, Higher levels means worse.

SECONDARY OUTCOMES:
Gingival Index | 30 days
  Check the biofilm as Ainano & Bay 1975 index, Higher levels means worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal Fluminense, Nova Friburgo, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No